CLINICAL TRIAL: NCT06398522
Title: Dietary Supplementation With Butyrate in Individuals With Liver Steatosis and Metabolic Syndrome: a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Dietary Supplementation With Butyrate in Individuals With Liver Steatosis and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Prof. Dr., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: But_17
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: NAFLD; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome | interventions — Food; gluconic acid; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food for special medical purposes (Active Comparator): Food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3
  Interventions: Dietary Supplement: Food for special medical purposes with calcium butyrate, zinc gluconate and vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food for special medical purposes with calcium butyrate, zinc gluconate and vitamin D3 — Food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3
  Arms: Food for special medical purposes
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This was a double-blind, randomized, placebo-controlled clinical study aiming to assess the effect of a food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3 on liver steatosis in individuals with NAFLD and metabolic syndrome

ELIGIBILITY:
Inclusion criteria:

* 40-75 years of age
* Caucasian ethnicity
* NAFLD
* Metabolic Syndrome

Exclusion criteria:

* acute and chronic gastrointestinal disorder not controlled by stable treatment since at least 3 months
* serious or disabling diseases (e.g. severe organ failure, malignancy or dementia)
* obesity (body mass index (BMI)> 30 Kg/m2)
* type 1 and 2 diabetes
* alcoholism
* pregnancy and breastfeeding
* any medical or surgical condition making complex or inconstant the adhesion to the study protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Effect on Fatty Liver Index | 3 months
  We evaluated the effect on Fatty Liver Index (FLI) of 3-month assumption of a food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3, compared to either baseline and placebo

SECONDARY OUTCOMES:
Effect on Hepatic Steatosis Index | 3 months
  We evaluated the effect on Hepatic Steatosis Index (HSI) of 3-month assumption of a food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3, compared to either baseline and placebo
Effect on Lipid Accumulation Product | 3 months
  We evaluated the effect on Lipid Accumulation Product (LAP) of 3-month assumption of a food for special medical purposes with functional release containing calcium butyrate, zinc gluconate and vitamin D3, compared to either baseline and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, BO, Italy